CLINICAL TRIAL: NCT02122380
Title: The Effect of Dipeptidyl Peptidase 4 Inhibition on Growth Hormone Secretion in Women With Polycystic Ovarian Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jessica Koch Devin, Principal Investigator, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 131969; K23HL119602-01A1 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-24 (Estimated); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Growth Hormone; Dipeptidyl Peptidase 4; Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin, then Placebo (Experimental): Sitagliptin 100 mg by mouth daily for 30 days followed by Placebo daily for 30 days
  Interventions: Drug: Sitagliptin; Drug: Placebo
- Placebo, then Sitagliptin (Experimental): Placebo daily for 30 days followed by Sitagliptin 100 mg daily for 30 days
  Interventions: Drug: Sitagliptin; Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg by mouth daily for 30 Days
  Other Names: Januvia
Drug: Placebo — 1 placebo pill by mouth per day for 30 days

SUMMARY:
Adults with abdominal obesity are at high risk for cardiovascular disease and also exhibit diminished growth hormone (GH) secretion; the latter further contributes to the development of visceral adiposity, impaired fibrinolysis and inflammation.Growth hormone releasing hormone (GHRH), the primary stimulus for endogenous GH secretion, is a substrate of dipeptidyl peptidase 4 (DPP4); inhibition of DPP4 with the currently available anti-diabetic therapy, sitagliptin, may therefore increase GH secretion by decreasing the degradation of GHRH. The proposed research will test the hypothesis that chronic sitagliptin therapy will enhance GH secretion and vascular function while improving glucose tolerance in patients with impaired GH secretion who are at risk for the development of diabetes mellitus and cardiovascular disease, specifically obese women with polycystic ovary syndrome.

DETAILED DESCRIPTION:
Thirty-four obese (BMI ≥ 30 kg/m2) females (18-40 years old) with polycystic ovarian syndrome (PCOS) will participate in this randomized, double-blind, placebo-controlled crossover study. The use of oral contraceptives or metformin will be discontinued at least 30 days prior. In females experiencing monthly cycles, the outpatient visit will take place during the mid-luteal phase of the participant's menstrual cycle and the inpatient visit will take place during the late follicular phase.

Subjects will be randomized to treatment order (sitagliptin 100 mg daily vs placebo) using a block randomization algorithm with a block size of two. The dose of sitagliptin was chosen as it is currently the FDA-recommended dose of sitagliptin for type 2 diabetic patients with unimpaired renal function. Subjects will receive standardized dietary counseling throughout the study; visits will be standardized to the menstrual cycle when possible. Subjects will take each therapy for one month; a minimum one month wash-out will separate study treatments. Side effects and compliance with study medication will be assessed at each visit in the clinical research center (CRC).

Each subject will undergo one outpatient visit and one inpatient visit during each treatment. On each study day, subjects will report fasting to the CRC in the morning having abstained from exercise that morning. On each study day, subjects will receive an intravenous catheter. Subjects will undergo an oral glucose tolerance test (OGTT) during the outpatient study visit. During the inpatient study visit, endothelium-dependent and -independent vasodilation will be assessed using flow-mediated dilation technique with ultrasound. Standardized meals will be provided at lunch and dinner. Body composition will be determined in the afternoon. At 8 PM overnight frequent sampling for venous GH will begin every 10 minutes for 12 hours to determine overnight GH secretion.

ELIGIBILITY:
Inclusion Criteria:

* Females, age 18-40 years
* BMI ≥ 30 kg/m2
* Diagnosis of polycystic ovary syndrome defined by 2003 Rotterdam criteria as meeting two out of the three below criteria :

  * Oligomenorrhea or amenorrhea
  * clinical or biochemical evidence of hyperandrogenism (hirsutism and/or documented upper normal or elevated serum testosterone in the absence of exogenous hormone therapy or Metformin)
  * documented history of polycystic ovaries on ultrasound examination

Exclusion Criteria:

* Smoking
* Type 1 or Type 2 Diabetes Mellitus, as defined by a fasting glucose of 126 mg/dL or greater at the time of screening visit or the use of anti-diabetic medication
* Hypertension, as defined by an untreated seated systolic blood pressure (SBP) greater than 150 mmHg and/or an untreated diastolic blood pressure (DBP) greater than 95 mmHg at the time of screening visit or the use of anti-hypertensive medication
* History of reported or recorded hypoglycemia (plasma glucose < 70 mg/dL)
* Pregnancy and/or Breast-Feeding (Negative serum pregnancy test will be confirmed at screening visit and every study visit.)
* Surgical menopause, defined as s/p total hysterectomy including bilateral salpingo-oophorectomy
* Use of transdermal or oral contraceptive therapy. The use of these contraceptives must be discontinued at least 8 weeks prior to study initiation.
* The use of insulin sensitizers, specifically Metformin or thiazolidinediones must be discontinued 8 weeks prior to study initiation.
* Anemia defined as hematocrit <35% at screening visit
* Cardiovascular or cerebrovascular disease, including history of myocardial infarction, history of congestive heart failure, history of stroke
* Pulmonary Hypertension
* Abnormal thyroid hormone levels (TSH), prolactin, or morning 17 hydroxyprogesterone at the time of screening visit
* Impaired renal function, defined as estimated glomerular filtration rate (eGFR) <60
* Impaired hepatic function (AST or ALT > 2 X upper limit of normal range)
* Treatment with an investigational drug in the 1 month preceding the study
* Allergy to any of the medications used in this protocol
* Regular work of a night-shift or unusual schedule which may disrupt circadian rhythm.
* Personal or Family History (defined as first degree relative) of Pancreatic Cancer
* Personal history of Pancreatitis or known pancreatic lesions
* Coagulopathy as defined by history
* Regular NSAID use, including but not limited to, naproxen, ibuprofen, and aspirin
* Mental conditions rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* Any underlying or acute disease requiring regular medication that could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-02; Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Devin, MD MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Devin JK, Nian H, Celedonio JE, Wright P, Brown NJ. Sitagliptin Decreases Visceral Fat and Blood Glucose in Women With Polycystic Ovarian Syndrome. J Clin Endocrinol Metab. 2020 Jan 1;105(1):136-51. doi: 10.1210/clinem/dgz028. PMID 31529097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 patients were screened for eligibility at Vanderbilt University Medical Center.
Pre-assignment Details: 23 out of 55 participants were randomized. Of those not randomized, 23 were did not meet inclusion criteria and 9 declined to participate.
Groups:
- Sitagliptin Then Placebo: Participants first received sitagliptin 100 mg by mouth daily for 30 days. After a washout period of 8 weeks, then then received Placebo daily for 30 days
- Placebo Then Sitagliptin: Participants first received Placebo daily for 30 days. After a washout period of 8 weeks, they then received Sitagliptin 100 mg daily for 30 days
Period: First Intervention (30 Days)
Arm/Group | Sitagliptin Then Placebo | Placebo Then Sitagliptin
Started | 11 | 12
Completed | 10 | 11
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Period: Washout (8 Weeks)
Arm/Group | Sitagliptin Then Placebo | Placebo Then Sitagliptin
Started | 10 | 11
Completed | 9 | 9
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — No Longer Met Inclusion Criteria | 0 | 2
Period: Second Intervention (30 Days)
Arm/Group | Sitagliptin Then Placebo | Placebo Then Sitagliptin
Started | 9 | 9
Completed | 9 | 7
Not Completed | 0 | 2
Not completed — 2 did not complete all of inpatient day | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants randomized to an intervention are included.
Groups:
- Sitagliptin Then Placebo: Participants first received sitagliptin 100 mg by mouth daily for 30 days. After an 8 week washout period, they then received Placebo daily for 30 days.
- Placebo Then Sitagliptin: Participants first received Placebo daily for 30 days. After an 8 week washout period, they then received Sitagliptin 100 mg daily for 30 days.
- Total: Total of all reporting groups
Arm/Group | Sitagliptin Then Placebo | Placebo Then Sitagliptin | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (4.3) | 30.3 (4.3) | 30.3 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Only Females were included in this study because Polycystic Ovarian Syndrome is a disorder limited to women.
  Participants
    Female | 11 | 12 | 23
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Overnight Growth Hormone Levels
Description: Growth hormone levels were determined every 10 minutes from 8 PM until 8 AM during the inpatient visit on the last day of each treatment. A mean of the GH levels was calculated for each participant, and then the value from each participant was averaged across all participants.
Time Frame: At completion of 30 days of placebo treatment and at completion of 30 days of sitagliptin treatment; every 10 minutes from 8 PM until 8 AM.
Population: All participants who received both interventions and completed both inpatient visits were included in the analysis. (1 participant was unable to complete their 2nd inpatient visit due to a family emergency. A 2nd participant was unable to complete the overnight portion of the inpatient visit due to illness in a family member.)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Placebo: Participants who received Placebo tablet each morning in either the first 30 days or last 30 days of the study.
- Sitagliptin: Participants who received Sitagliptin 100 mg daily each morning in either the first 30 days or last 30 days of the study.
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 16 | 16
ng/mL | 0.85 (0.54) | 0.84 (0.51)
Statistical Analysis 1: Comparison: Placebo vs Sitagliptin; Null hypothesis is that there was no difference in change of mean growth hormone (GH) levels between sitagliptin and placebo. The test was performed with a significance level of 0.05 (two sided). A sample size of 16 participants was needed to provide 93% power to detect a difference in GH means of 0.5 mcg/L; Test type: Superiority; p = 0.918, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Early Insulin Secretion During Oral Glucose Tolerance Test
Description: Oral glucose tolerance testing was performed with 75 grams of glucose solution. Baseline venous blood samples of insulin were obtained prior to ingestion of oral glucose solution (time 0). Insulin levels were then obtained through a peripheral IV line every 15 minutes for 270 minutes after glucose solution is swallowed. Early insulin secretion was determined by calculating area under the curve using data (i.e. insulin levels) obtained at baseline (time 0), 15 minutes and 30 minutes.
Time Frame: During Outpatient Visit (after 2 weeks of therapy) during placebo and sitagliptin treatment periods. Insulin levels were obtained at time 0, 15 and 30 minutes following 75 gram glucose ingestion.
Population: All participants who received both interventions and completed both outpatient study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: microU*minutes/mL
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 18 | 18
microU*minutes/mL | 1522.1 (792.3) | 1871.3 (843.6)
Statistical Analysis 1: Comparison: Placebo vs Sitagliptin; Null hypothesis is that there was no difference in change of early insulin secretion between sitagliptin and placebo. The test was performed with a significance level of 0.05 (two sided); Test type: Superiority; p = 0.054, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Area Under the Curve (AUC) for Blood Glucoses During 75 Gram Oral Glucose Tolerance Test
Description: Oral glucose tolerance testing was performed with 75 grams of glucose solution. Baseline blood glucose was obtained prior to ingestion of oral glucose solution (time 0). Blood glucose levels were then obtained through a peripheral IV line every 15 minutes from timepoint 0 until 120 minutes to calculate the area under the curve.
Time Frame: During Outpatient Visit (after 2 weeks of therapy) during placebo and sitagliptin treatment periods. Every 15 minutes from time 0 to 120 minutes after oral glucose ingestion.
Population: All participants who received both interventions and completed both outpatient study visits were included in analysis.
Measure: Mean (Standard Deviation); unit: mg*minutes/dL
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 18 | 18
mg*minutes/dL | 15353.8 (2708.6) | 13877.5 (2486.3)
Statistical Analysis 1: Comparison: Placebo vs Sitagliptin; Null hypothesis is that there was no difference in blood glucose levels between sitagliptin and placebo. The test was performed with a significance level of 0.05 (two sided); Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Visceral Adipose Tissue
Description: During the inpatient visit of each treatment (placebo and sitagliptin), visceral adipose tissue was determined by a certified densitometrist using dual-energy x-ray absorptiometry with enCore software (v. 13.6)
Time Frame: At completion of 30 days of placebo treatment and at completion of 30 days of sitagliptin treatment.
Population: All participants who received both interventions and completed all study protocols during the daytime portion of the inpatient visits were included in the analysis. (1 participant was unable to complete their 2nd inpatient visit due to a family emergency.)
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Sitagliptin: Participants who received Sitagliptin 100 mg each morning in either the first 30 days or last 30 days of the study.
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 17 | 17
grams | 1141.9 (700.7) | 1055.1 (710.1)
Statistical Analysis 1: Comparison: Placebo vs Sitagliptin; Null hypothesis is that there was no difference in the mass of visceral adipose tissue after sitagliptin vs. placebo. The test was performed with a significance level of 0.05 (two sided); Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Vascular Function (Endothelium-dependent Vasodilation)
Description: Endothelium-dependent vasodilation was evaluated by measuring the diameter of the brachial artery under basal (i.e. rest) condition and during reactive hyperemia. The percentage change in diameter (i.e. endothelium-dependent vasodilation) was calculated as percent change=[(peak diameter-baseline diameter)/baseline diameter]*100. Endothelium-dependent vasodilation was determined twice during the study: at completion of 30 days of placebo treatment and at completion of 30 days of sitagliptin treatment.
Time Frame: Vascular function was determined by measuring brachial artery diameter at rest and during reactive hyperemia and calculating percent change. This was determined after 30 days of placebo treatment and after 30 days of sitagliptin treatment.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 17 | 17
percent change | 13.63 (5.27) | 13.00 (5.34)
Statistical Analysis 1: Comparison: Placebo vs Sitagliptin; Null hypothesis is that there was no difference in vascular function between sitagliptin and placebo treatments. The test was performed with a significance level of 0.05 (two sided); Test type: Superiority; p = 0.943, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 30 days for each intervention.
Description: Safety population included all participants who received at least one dose of intervention.
Groups:
- Sitagliptin: Participants received Sitagliptin 100 mg by mouth daily for up to 30 days.
- Placebo: Participants received Placebo daily for up to 30 days.
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/21
Other Adverse Events (participants affected / at risk) | 5/20 | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=20) | Placebo (N=21)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=20) | Placebo (N=21)
Abdominal Pain, Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Shingles Infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT02122380/Prot_SAP_000.pdf